CLINICAL TRIAL: NCT04265105
Title: A Pilot Randomised Controlled Superiority Trial of Fluticasone-Vilanterol Once Daily Dose for the Treatment of Mild Asthma in Adults
Brief Title: Fluticasone-Vilanterol Once Daily Dose for the Treatment of Mild Asthma in Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Responsible Party: Principal Investigator, Dr Ghufran Jassim, Associate professor, Royal College of Surgeons in Ireland - Medical University of Bahrain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCSIBahrain
Record Dates: First submitted 2020-01-14; First posted 2020-02-11 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: asthma; fluticasone; LABA; fluticasone-vilanterol; Long acting Beta agonist
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate-vilanterol trifenatate; Reference Standards; Standard of Care

STUDY DESIGN:
Intervention Model Description: Investigators will compare the superiority of effectiveness and safety of fluticasone-vilanterol versus usual care. In this study, there is a random allocation of participants to usual care (Any ICS or SABA combination) or fluticasone-vilanterol single daily use for the relief of symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (Active Comparator): Short acting beta agonist or inhaled corticosteroids
  Interventions: Drug: Standard Preparation
- fluticasone-vilanterol (Experimental): LABA-ICS A combination of Long acting beta agonist and inhaled corticosteroid
  Interventions: Drug: fluticasone-vilanterol

INTERVENTIONS:
Drug: fluticasone-vilanterol — LABA-ICS combination Inhaled Long acting Beta agonist and inhaled corticosteroid
  Arms: fluticasone-vilanterol
Drug: Standard Preparation — inhaled SABA or Inhaled corticosteroid
  Other Names: standard of care
  Arms: standard of care

SUMMARY:
Investigators will test the superiority of Superiority Trial of Fluticasone-Vilanterol as needed in mild asthma compared to standard of care

DETAILED DESCRIPTION:
single centre randomised control trial with the aim of comparing the superiority of effectiveness and safety of fluticasone-vilanterol versus usual care. In this study there is random allocation of participants to usual care (Any ICS or SABA combination) or fluticasone-vilanterol daily single dose for the relief of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 75 years old with a diagnosis of mild asthma attending the participating primary health care centres in Bahrain, being managed with usual care (SABA or ICS and SABA combination) and no other medications

Exclusion Criteria:

* Health centre medical record or self-reported use of LABA, leukotriene receptor agonist, theophylline, anticholinergic agent, oral corticosteroids for regular maintenance therapy in 3 months before entry to the trial. [NB. nasal corticosteroid is permitted

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Number of asthma exacerbations | 32 weeks/8 months
  measured by asking the participants about Hospital admission with asthma/ Visit to ED with Asthma and receiving treatment with nebulizer and/ or any corticosteroids (IV, IM, PO or neb)/ Home use of nebulizer and/or corticosteroids (IV, IM, oral or nebulized). treatment with nebulizer and/ or any corticosteroids (IV, IM, PO or neb)/ Home use of nebulizer and/or corticosteroids (IV, IM, oral or nebulized)
Change in Asthma Control Score | baseline, 8 months
  measured by the 7 item asthma control questionnaire. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control.

SECONDARY OUTCOMES:
Change in Asthma Quality of life score | baseline, 8 months
  Measured using a 32 item questionnaire Scores range 1-7, with higher scores indicating better quality of life. a minimal important within-subject change in an AQLQ subscale or overall scale score is 0.5, with changes of 1.0 considered moderate and changes of 2.0 considered large

CONTACTS AND LOCATIONS:
Locations (1):
- RCSI Bahrain, Al Muharraq, Busaiteen, Bahrain

IPD SHARING:
Plan to Share IPD: No
Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 3 years after study completion (last patient, last visit). A label stating the date after which the documents can be destroyed will be placed on the inside front cover of the case notes of trial participants.Monitoring, audits, and REC review will be permitted and provide direct access to source data and documents. The Lead PI and the researcher assigned by her will have access to the stored data. Only the CRCs and Lead PI working on this study will be eligible to obtain the data from the participants during data collection visits.